CLINICAL TRIAL: NCT07122856
Title: Predictive Factors for Initial MMSE Score and Rapid Decline in Alzheimer's Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0114_NEUROLOGIE_TARGET MMSE
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Mini-Mental State Examination; Cognitive Dysfunction; Neuropsychological Tests; Caregivers
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks at people with Alzheimer's disease to find out which factors are linked to their initial score on the Mini-Mental State Examination (MMSE) and which factors may predict a fast decline in their score over 12 months. Researchers will review medical records from patients seen at the Memory Clinic of Gonesse Hospital and analyze information such as age, education, medical history, nutrition, mood, and caregiver burden. The goal is to better understand what influences early cognitive performance and how quickly it changes, to help improve patient care and planning.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Alzheimer's disease according to NIAA 2018 or IWG 2021 criteria
* At least two MMSE evaluations spaced 12 months apart
* Follow-up at the Memory Clinic of CH Gonesse

Exclusion Criteria:

* Presence of other neurodegenerative diseases (e.g., Frontotemporal Dementia, Multiple System Atrophy, Vascular Dementia, LATE)
* Patient has moved out of the study area (outside the CH Gonesse territory)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of all patients who attended the Memory Clinic at CH Gonesse between July 2023 and July 2025. From this group, participants will be selected if they have a confirmed diagnosis of Alzheimer's disease (based on NIAA 2018 or IWG 2021 criteria) and have undergone at least two MMSE assessments spaced 12 months apart. Data will be extracted from medical records and registries within this hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in MMSE Score Over 12 Months - measured as either a decrease of ≥3 points on the Mini-Mental State Examination [MeSH] or patient institutionalization within 12 months. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Gonesse, Gonesse, France, France